CLINICAL TRIAL: NCT06400446
Title: The Effect of Kangaroo Care on Vital Signs of Infants After Cardiac Surgery
Brief Title: The Effect of Kangaroo Care After Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ISU-23-259
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Infant ALL
Keywords: Kangaroo care; Infant; Cardiac surgery; Vital signs
MeSH Terms: interventions — Standard of Care; Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (standard care) (Other): The babies in this group will receive the standard care of the unit.
  Interventions: Other: Standard care
- Experimental group (Kangaroo care) (Experimental): Kangaroo care will be applied to the experimental group for seven days.
  Interventions: Other: Kangaroo care

INTERVENTIONS:
Other: Standard care — The babies in this group will receive the standard care of the unit. The vital signs and pain scores of the babies will be recorded before the mother's visit for seven days. The vital signs and pain scores of the infants who received the standard care of the unit during one hour, which is the time of the mother's visit, will be recorded every 15 minutes for a total of 4 times. The vital signs and pain scores of the infant will be recorded in the first 15 minutes after the mother's visit.
  Arms: Control group (standard care)
Other: Kangaroo care — Kangaroo care will be applied to the experimental group for seven days. Kangaroo care will be started for the babies in the intervention group when the baby is extubated, when the baby starts oral feeding and when the chest incision is closed. Consistent with previous research, mothers will provide skin-to-skin contact for at least 1 hour per day for seven days, starting immediately after feeding. The vital signs and pain scores of the babies will be recorded during the kangaroo care of the mother for seven days. During the kangaroo care, vital signs and pain scores of the infants will be recorded every 15 minutes for a total of 4 times. The vital signs and pain scores of the infant will be recorded in the first 15 minutes after the mother's visit.
  Arms: Experimental group (Kangaroo care)

SUMMARY:
The aim of this study was to investigate the effects of kangaroo care on the vital signs of infants undergoing cardiac surgery.

Hypothesis 1 (H1): Oxygen saturation levels of babies who are given kangaroo care are higher than babies who are not given kangaroo care.

Hypothesis 2 (H2): The peak heart rate of infants who receive kangaroo care is lower than infants who do not receive kangaroo care.

Hypothesis 3 (H3): The respiratory rate of infants who receive kangaroo care is lower than infants who do not receive kangaroo care.

Hypothesis 4 (H4): The arterial blood pressure of infants who receive kangaroo care is lower than infants who do not receive kangaroo care.

Hypothesis 5 (H5): The pain score of infants who received kangaroo care is lower than infants who did not receive kangaroo care.

DETAILED DESCRIPTION:
Kangaroo care has been found to be a feasible intervention before and after cardiac surgery to support infants with congenital heart disease, but it has been stated that formal standards and procedures need to be developed to transform kangaroo care into practice. Skin-to-skin contact is a low-cost, low-risk intervention that supports comfort and contributes to physiological stability in infants before and after neonatal cardiac surgery. It positively affects the pain level of infants. Clinical studies on the application of kangaroo mother care on infants undergoing cardiac surgery are limited in the literature.

ELIGIBILITY:
Inclusion Criteria:

* The gestational week of the infant is greater than 37 weeks
* Cardiac surgery operation within the first 30 days of life
* The infant's chest incision is closed

Exclusion Criteria:

* The infant has non-cardiac congenital defects or syndrome
* Intubation of the infant

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Change in oxygen saturation | Data will be collected immediately before care is given, at 15 minutes during care, and at 15 minutes after care is given. The change in these time intervals will be evaluated.
  Oxygen saturation will be monitored.
Change in heart rate | Data will be collected immediately before care is given, at 15 minutes during care, and at 15 minutes after care is given. The change in these time intervals will be evaluated.
  Heart rate will be monitored.
Change in respiratory rate | Data will be collected immediately before care is given, at 15 minutes during care, and at 15 minutes after care is given. The change in these time intervals will be evaluated.
  Respiratory rate will be monitored.
Change in blood pressure | Data will be collected immediately before care is given, at 15 minutes during care, and at 15 minutes after care is given. The change in these time intervals will be evaluated.
  Blood pressure will be monitored.
Change in level of pain | Data will be collected immediately before care is given, at 15 minutes during care, and at 15 minutes after care is given. The change in these time intervals will be evaluated.
  The infants' pain level will be measured using the CRIES(Crying, Requires O2, Increased vital signs,Expression, Sleepless). The scale is used in the evaluation of postoperative pain in premature babies (between 32-36 weeks of gestation) and postoperative pain. Starting from the thirty-second gestational week, it is preferred in neonates and children between 6 months, especially in intensive care units.The Scale was developed by Krechel & Bildner, 1995. Crying status, oxygen saturation, heart rate and/or blood pressure, facial expression and sleep status are the parameters used in the evaluation. Each parameter is scored out of two; a score of 3-4 indicates mild to moderate pain; values of five and above indicate severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Cengizli, Nurse, Principal Investigator — Istanbul Health Sciences University Mehmet Akif Ersoy Chest Heart and Vascular Surgery Training and Research Hospital Paediatric Cardiovascular Surgery Intensive Care Unit
Locations (1):
- Selvinaz Albayrak, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Solaz-Garcia A, Lara-Canton I, Pinilla-Gonzalez A, Montejano-Lozoya R, Gimeno-Navarro A, Sanchez-Illana A, Marco-Pinol A, Vento M, Saenz-Gonzalez P. Impact of Kangaroo Care on Premature Infants' Oxygenation: Systematic Review. Neonatology. 2022;119(5):537-546. doi: 10.1159/000525014. Epub 2022 Jun 22. PMID 35732143
- [Result] Kelley-Quon LI, Kenney BD, Bartman T, Thomas R, Robinson V, Nwomeh BC, Bapat R. Safety and feasibility of skin-to-skin care for surgical infants: A quality improvement project. J Pediatr Surg. 2019 Nov;54(11):2428-2434. doi: 10.1016/j.jpedsurg.2019.02.016. Epub 2019 Feb 28. PMID 30879741
- [Result] Lisanti AJ, Vittner D, Medoff-Cooper B, Fogel J, Wernovsky G, Butler S. Individualized Family-Centered Developmental Care: An Essential Model to Address the Unique Needs of Infants With Congenital Heart Disease. J Cardiovasc Nurs. 2019 Jan/Feb;34(1):85-93. doi: 10.1097/JCN.0000000000000546. PMID 30303895